CLINICAL TRIAL: NCT01074684
Title: Defining Predictive Factors of Clinical, Laboratory and Imaging Criteria Routinely Used in the Diagnosis of Thyroid Cancer: Observational, Prospective Multicentered Study
Brief Title: Predictive Factors of Clinical, Laboratory and Imaging Findings Routinely Used in Diagnosing Thyroid Cancer
Acronym: TIR-2009-01
Status: Completed | Type: Observational
Sponsor: National Cancer Institute, Naples (Other)
Responsible Party: Sponsor
Other Study IDs: TIR-2009-01
Record Dates: First submitted 2010-02-23; First posted 2010-02-24 (Estimated); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Thyroid Cancer
Keywords: diagnosis; nodules; fine needle aspiration
MeSH Terms: conditions — Thyroid Neoplasms; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to describe the correlation between the cytohistology exam of patients undergoing thyroid surgery, and the predictive values of: suspicious clinical findings, preoperative thyroid imaging, and the incidence of thyroid cancer in cytologically negative nodes.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients presenting for thyroid disease (palpable nodules)
* Indication for surgery
* Age > 18 years
* Signed informed consent for surgery
* Signed informed consent for data collection

Exclusion Criteria:

* Concurrent condition that contraindicates surgery
* Clinical or radiologic evidence of locally advanced tumor
* Clinical or radiologic evidence of metastatic lymph nodes or distant metastases
* Nonpalpable nodes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients with palpable thyroid nodules with indication for surgery (positive cytology, 2 consecutive inconclusive cytologies, or negative cytology with at least 2 of the following: previous exposure to neck radiation, calcitonin greater than twice normal values, positive pentagastrin test, or irregular margins or hypoechogenicity on ultrasound.
Sampling Method: Non-Probability Sample
Enrollment: 959 (Actual)
Dates: Start 2010-01; Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
positive predictive value of preoperative suspicious clinical, laboratory and imaging findings | at baseline

CONTACTS AND LOCATIONS:
Overall Officials: Luciano Pezzulo, M.D., Principal Investigator — National Cancer Institute, Naples; Maria Grazia Chiofalo, M.D., Principal Investigator — National Cancer Institute, Naples; Massimo Di Maio, M.D., Principal Investigator — National Cancer Institute, Naples; Francesco Perrone, M.D., Ph.D., Principal Investigator — National Cancer Institute, Naples
Locations (8):
- Italy (8):
  - Università di Cagliari, Cagliari
  - Azienda Ospedaliera Unviersitaria Careggi - Firenze, Florence
  - ASL TO/4 Ospedale di Ivrea, Ivrea
  - Istituto Nazionale dei Tumori, Napoli
  - Azienda Ospedaliera Universitaria di Padova, Padua
  - Università Cattolica del Sacro Cuore di Roma Policlinico Gemelli, Roma
  - Ospedale di Taormina, Taormina
  - Università degli studi di Perugia - Sede di Terni, Terni